CLINICAL TRIAL: NCT01052662
Title: Memantine-enhanced Buprenorphine Treatment for Opioid-dependent Young Adults
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: University of Massachusetts, Worcester (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Principal Investigator, Gerardo Gonzalez, Principal Investigator, University of Massachusetts, Worcester
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: H-13261; 1R01DA027138-01 (NIH)
Record Dates: First submitted 2010-01-18; First posted 2010-01-20 (Estimated); Results first posted 2015-03-06 (Estimated); Last update posted 2015-04-01 (Estimated); Status verified 2015-03

CONDITIONS: Opioid Dependence
Keywords: Drug Abuse
MeSH Terms: conditions — Opioid-Related Disorders; Substance-Related Disorders | interventions — Memantine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Memantine 30mg/day + Buprenorphine (Experimental): Participants were inducted onto buprenorphine/naloxone sublingual tablets during the first week of study participation. The dose was titrated from bup/nal 8mg to bup/nal 16mg in three days where it will remain until the last day of week 8. The 7-day discontinuation of buprenorphine-naloxone on week 9 was 12mg, 10mg, 8mg, 6mg, 4mg, 2mg, 2mg and stopped.
  Memantine 5mg in the morning was started on week 2. The dose was titrated on a twice a day schedule until the target dose of 30 mg/day was achieved by week 4. The medication was discontinued over a one-week period on week 13. Patients received a 7-day supply of their medication each week.
  Interventions: Drug: Memantine
- Memantine 15mg/day + Buprenorphine (Experimental): Participants were inducted onto buprenorphine/naloxone sublingual tablets during the first week of study participation. The dose was titrated from bup/nal 8mg to bup/nal 16mg in three days where it will remain until the last day of week 8. The 7-day discontinuation of buprenorphine-naloxone on week 9 was 12mg, 10mg, 8mg, 6mg, 4mg, 2mg, 2mg and stopped.
  Memantine 5mg in the morning was started on week 2. The dose was titrated on a twice a day schedule until the target dose of 15 mg/day was achieved by week 4. The medication was discontinued over a one-week period on week 13. Patients received a 7-day supply of their medication each week.
  Interventions: Drug: Memantine
- Memantine 0mg/day + Buprenorphine (Placebo Comparator): Participants were inducted onto buprenorphine/naloxone sublingual tablets during the first week of study participation. The dose was titrated from bup/nal 8mg to bup/nal 16mg in three days where it will remain until the last day of week 8. The 7-day discontinuation of buprenorphine-naloxone on week 9 was 12mg, 10mg, 8mg, 6mg, 4mg, 2mg, 2mg and stopped.
  Matching placebo capsule was started on week 2. The placebo capsules were given on a twice a day schedule until week 12 and then discontinued over a one-week period on week 13. Patients received a 7-day supply of their medication each week.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Memantine — 30mg/day Memantine orally everyday for 12 weeks
  Arms: Memantine 30mg/day + Buprenorphine
Drug: Memantine — 15 mg/day Memantine orally everyday for 12 weeks
  Arms: Memantine 15mg/day + Buprenorphine
Drug: Placebo — Placebo orally everyday for 12 weeks
  Arms: Memantine 0mg/day + Buprenorphine

SUMMARY:
The purpose of this study is to examine the effect of memantine and buprenorphine on opioid abusing behavior, to determine the effect of memantine and buprenorphine on early relapse and to evaluate the tolerability of memantine co-administrated with buprenorphine. The study seeks to determine if combined treatment of memantine and buprenorphine may provide shorter-term treatment for opioid dependence.

DETAILED DESCRIPTION:
Opiate dependence is an increasing problem among young adults (18-25 years old) whose rates of current use of illicit drugs are generally high (19.7 %)according to data from the 2007 National Survey on Drug Use & Health (Substance Abuse and Mental Health Services Administration 2008). Young adults start using heroin around this age range, and more recently have had increasing rates of prescription-type drug use. Given that young adults with opiate dependence who are seeking treatment are relatively treatment naïve, have a shorter period of addiction, and are more likely to choose buprenorphine over methadone, developing short-term buprenorphine treatment alternatives to long-term methadone agonist treatment is needed.

ELIGIBILITY:
Inclusion Criteria:

* Men and women between 18-25 years old
* Opioid dependence as evidenced by signs of opiate withdrawal, self-reported history of opioid dependence for a consecutive 12 month period and positive urine for opioids

Exclusion Criteria:

* Current diagnosis of other drug or alcohol dependence (other than opiates, cannabis or tobacco)
* Serious medical illness (e.g. major cardiovascular, renal, endocrine, hepatic disorder)
* Current serious psychiatric illness or history of psychosis, schizophrenia, bipolar type I disorder and participants with suicidal or homicidal thoughts
* Women who are pregnant, nursing or refuse to use a reliable form of birth control or refuse monthly pregnancy testing
* Screening liver function tests (SGOT or SGPT) greater than 3 times normal

Ages: 18 Years to 25 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 87 (Actual)
Dates: Start 2009-10; Primary Completion 2013-06 (Actual); Study Completion 2013-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Gerardo Gonzalez, M.D., Principal Investigator — University of Massachusetts, Worcester
Locations (1):
- University of Massachusetts Medical School, Worcester, Massachusetts, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment was done by newspaper advertising, referrals from the University of Massachusetts Addiction and Comorbidity Treatment Service (ACTS) and from community-based substance abuse clinics.
Pre-assignment Details: 229 individuals of the 354 persons who were interested in the study were assessed not eligible to participate. Of the 125 subjects that were screen over one week, only 87 subjects meet criteria for study participation. Reason for exclusion included: declined (N=22), psychiatric (N=6), other SUD (N=6), abnormal labs (N=3) and medical reason (N=1)
Groups:
- Memantine 30mg/Day + Buprenorphine: Participants were inducted onto buprenorphine/naloxone sublingual tablets during the first week of study participation. The dose was titrated from bup/nal 8mg to bup/nal 16mg in three days where it will remain until the last day of week 8. The 7-day discontinuation of buprenorphine-naloxone on week 9 was 12mg, 10mg, 8mg, 6mg, 4mg, 2mg, 2mg and stopped.
  Memantine 5mg in the morning was started on week 2. The dose was titrated on a twice a day schedule until the target dose of 30 mg/day was achieved by week 4. The medication was discontinued over a one-week period on week 13. Patients received a 7-day supply of their medication each week.
  Memantine: 30mg/day Memantine orally everyday for 12 weeks
- Memantine 15mg/Day + Buprenorphine: Participants were inducted onto buprenorphine/naloxone sublingual tablets during the first week of study participation. The dose was titrated from bup/nal 8mg to bup/nal 16mg in three days where it will remain until the last day of week 8. The 7-day discontinuation of buprenorphine-naloxone on week 9 was 12mg, 10mg, 8mg, 6mg, 4mg, 2mg, 2mg and stopped.
  Memantine 5mg in the morning was started on week 2. The dose was titrated on a twice a day schedule until the target dose of 15 mg/day was achieved by week 4. The medication was discontinued over a one-week period on week 13. Patients received a 7-day supply of their medication each week.
  Memantine: 15 mg/day Memantine orally everyday for 12 weeks
- Memantine 0mg/Day + Buprenorphine: Participants were inducted onto buprenorphine/naloxone sublingual tablets during the first week of study participation. The dose was titrated from bup/nal 8mg to bup/nal 16mg in three days where it will remain until the last day of week 8. The 7-day discontinuation of buprenorphine-naloxone on week 9 was 12mg, 10mg, 8mg, 6mg, 4mg, 2mg, 2mg and stopped.
  Matching placebo capsule was started on week 2. The placebo capsules were given on a twice a day schedule until week 12 and then discontinued over a one-week period on week 13. Patients received a 7-day supply of their medication each week.
  Placebo: Placebo orally everyday for 12 weeks
Period: Overall Study
Arm/Group | Memantine 30mg/Day + Buprenorphine | Memantine 15mg/Day + Buprenorphine | Memantine 0mg/Day + Buprenorphine
Started | 28 (1 subject excluded from Intent-to-treat sample for final analysis due to pharmacy issue.) | 27 (3 subjects excluded from Intent-to-treat sample for final analysis due to pharmacy issue) | 32 (3 subjects excluded from Intent-to-treat sample for final analysis due to pharmacy issue)
Stabilization Phase | 21 | 21 | 26
Discontinuation Phase | 6 | 5 | 10
Completed | 6 | 5 | 10
Not Completed | 22 | 22 | 22
Not completed — Lost to Follow-up | 15 | 13 | 18
Not completed — Withdrawal by Subject | 3 | 2 | 1
Not completed — Pharmacy issue | 1 | 3 | 3
Not completed — Adverse Event | 1 | 1 | 0
Not completed — Legal Problem | 2 | 0 | 0
Not completed — Administrative | 0 | 3 | 0

BASELINE CHARACTERISTICS:
Population: Intent-to-treat sample
Groups:
- Total: Total of all reporting groups
Arm/Group | Memantine 30mg/Day + Buprenorphine | Memantine 15mg/Day + Buprenorphine | Memantine 0mg/Day + Buprenorphine | Total
Number analyzed (Participants) | 27 | 24 | 29 | 80
Age, Continuous [Mean (Standard Deviation); unit: years] | 23 (1.9) | 22.4 (2) | 22.4 (2.1) | 22.6 (1.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8 | 10 | 9 | 27
  Male | 19 | 14 | 20 | 53
Race/Ethnicity, Customized [Number; unit: participants]
  Caucacian | 25 | 21 | 27 | 73
  Hispanic | 2 | 3 | 2 | 7
Region of Enrollment [Number; unit: participants]
  United States | 27 | 24 | 29 | 80
Opioid use [Number; unit: participants]
  Heroin use | 5 | 7 | 5 | 17
  Opioid analgesic use | 22 | 17 | 24 | 63
Years of opioid use [Mean (Standard Deviation); unit: years]
  Heroin use | 1.1 (2.5) | 1 (1.6) | 1.1 (2.3) | 1.08 (2.1)
  Opioid Analgesic use | 2.8 (2.1) | 2.9 (1.3) | 3.7 (2.2) | 3.2 (1.9)
Severity of Dependence Scale [Mean (Standard Deviation); unit: units on a scale] — Performed at screening, we used this scale for urn randomization based on the severity of opiate dependence score. This instrument has 5 questions that are scored on a four-point scale from 0 ( never/almost never or not difficult) to 3 (always/nearly always or impossible). Overall scores range from 0 to 15, with scores above 10 indicating high severity.
  units on a scale | 11.2 (2.1) | 11.7 (2.5) | 11.7 (2.5) | 11.5 (2.4)
Clinical Opiate Withdrawal Scale (COWS) [Mean (Standard Deviation); unit: units on a scale] — The COWS is an 11-item interviewer administered questionnaire designed to provide a description of signs and symptoms of opiate withdrawal that can be observed directly in the participant (e.g., sweating, runny nose, etc). Scores range from 0 to 36. Score 5-12 = Mild, 13-24 = Moderate, 25-36 = Moderately Severe and more than 36 = Severe Withdrawal.
  units on a scale | 10.4 (3.7) | 8.3 (2.8) | 9.1 (2.7) | 9.2 (3.1)
Heroin Craving Questionnaire - Short Form 14 (HCQ-SF-14) [Mean (Standard Deviation); unit: units on a scale] — The Heroin Craving Questionnaire - Short Form 14 (HCQ-SF-14) consists of 14 statements about the respondent's feelings and thoughts about using heroin as he or she is completing the questionnaire (i.e., right now). This instrument obtains a reflection of the respondent's general heroin craving. This instrument was modified to include craving for prescription opioids. Each item is scored on a scale ranging from 1 for "Strongly Disagree" to 7 for "Strongly Agree." The total score is the average of the sum all 14 items with range from 1 to 7 with higher score indicating worse craving.
  units on a scale | 4.2 (1.1) | 4.5 (1) | 4.3 (1) | 4.3 (1)
Center for Epidemiologic Studies Depression scale (CES-D) [Mean (Standard Deviation); unit: units on a scale] — CES-D is a 20-item self-report measure of depressive symptoms. CES-D was administered at intake and weekly. The range of scores is from 0 to 60, with higher scores reflecting increased depressive symptoms. The CES-D does not heavily depend on pathological items or somatic symptoms compared with other scales.
  units on a scale | 23.6 (9) | 20 (9.7) | 22.8 (11) | 22.4 (9.9)
Barratt Impulsivity Questionnaire [Mean (Standard Deviation); unit: units on a scale] — The Barratt Impulsivity Questionnaire is a brief, participant-administered 30-item, self-rating scale where participants answer questions regarding behavior and planning using a four-point scale (1= Rarely/Never, 2= Occasionally, 3= Often, 4= Almost always/Always) where the maximum overall impulsivity score is 120 indicating more impulsive and the minimum score is 30.
  units on a scale | 72.4 (10.9) | 70.4 (10.3) | 69.7 (12.7) | 70.8 (11.3)
Inhibitory Control (mean % error) [Mean (Standard Deviation); unit: mean percentage of error (prosaccade)] — Antisaccade Task: Participants view a computer screen displaying two placeholder outline boxes on either side of a fixation cross. Subjects are instructed to look away from the go signal when it appears inside one of the placeholder boxes. For each trial, the first saccade that follows the go signal will be labeled an impulsivity error (i.e., a prosaccade) if it lands on the box containing the go signal and a correct response (i.e., an antisaccade) if it lands in the goal box. This task is an excellent measure of the control over impulsive behavior with higher scores indicating worse control.
  mean percentage of error (prosaccade) | 0.24 (0.2) | 0.2 (0.11) | 0.2 (0.17) | 0.21 (0.17)

OUTCOME MEASURES:

1. Primary Outcome: Change of Opioid Use From Week 1 to 13
Description: The primary outcome variable was the change from baseline of the mean proportion of weekly opioid use assessed by self-reported days of use and/or positive urine drug screen during the previous week using the time-line followed-back method (TLFB) . A positive urine counted as 1, as did each self-reported day of use. Each participants total was divided by 8. Mean proportion by group were calculated by averaging the proportions across participants in that group.
Time Frame: Weekly from week 1 to 13
Population: 80 subjects intent-to-treat.
Measure: Mean (Standard Error); unit: Mean Proportion of Opioid Use in Week 13
Arm/Group | Memantine 30mg/Day + Buprenorphine | Memantine 15mg/Day + Buprenorphine | Memantine 0mg/Day + Buprenorphine
Number analyzed (Participants) | 27 | 24 | 29
Mean Proportion of Opioid Use in Week 13 | 0.00 (0.0) | 0.27 (0.10) | 0.39 (0.14)
Statistical Analysis 1: Comparison: Memantine 30mg/Day + Buprenorphine vs Memantine 15mg/Day + Buprenorphine vs Memantine 0mg/Day + Buprenorphine; We modeled the mean proportion of weekly opioid use using a mixed-effect linear regression approach to assess the treatment effect, the time effect and the interaction of time x treatment effect while adjusting for the baseline mean proportion of weekly opioid use with baseline COWS, Addiction Severity Index (ASI) psychiatric and legal composite scores as covariates; Test type: Superiority or Other; p = 0.00874, Mixed Models Analysis; Slope = -0.00935, Standard Error of Mean 0.00356 — Z = -2.62209

2. Secondary Outcome: Treatment Retention
Description: Treatment retention during the stabilization period weeks 1 to 8 and after buprenorphine / naloxone discontinuation weeks 9 to 13.
Time Frame: Weekly
Population: Intent-treat-sample (ITT) that was inducted onto buprenorphine / naloxone and received one dose of study medication on week 2.
Measure: Mean (95% Confidence Interval); unit: weeks in treatment
Arm/Group | Memantine 30mg/Day + Buprenorphine | Memantine 15mg/Day + Buprenorphine | Memantine 0mg/Day + Buprenorphine
Number analyzed (Participants) | 27 | 24 | 29
weeks in treatment | 9.3 [8.3 to 10.2] | 9 [7.8 to 10.3] | 9.7 [8.6 to 10.6]
Statistical Analysis 1: Comparison: Memantine 30mg/Day + Buprenorphine vs Memantine 15mg/Day + Buprenorphine vs Memantine 0mg/Day + Buprenorphine; Test type: Superiority or Other; p = 0.64, Log Rank; Hazard Ratio, log = 0.87

3. Primary Outcome: Number of Participants Who Were Estimated to Have Survived as Assessed by Survival Curve of Relapse Rate After Achieving Complete Abstinence on Week 8
Description: Calculated survival curve from abstinence in Week 8 to first positive opioid urine screen or first reported relapse to opioid use to evaluate the effect of memantine on reducing early relapse and after rapid buprenorphine discontinuation on week 9. The last observation carried forward (LOCF) was used to perform our event survival analyses.
Time Frame: Weeks after buprenorphine discontinuation week 9
Population: Participants that achieved complete abstinence by self-report that was confirmed with negative urine toxicology at week 8.
Measure: Number; unit: participants
Arm/Group | Memantine 30mg/Day + Buprenorphine | Memantine 15mg/Day + Buprenorphine | Memantine 0mg/Day + Buprenorphine
Number analyzed (Participants) | 12 | 3 | 14
participants | 5 | 1 | 8
Statistical Analysis 1: Comparison: Memantine 30mg/Day + Buprenorphine vs Memantine 0mg/Day + Buprenorphine; Test type: Superiority or Other; p = 1.2, Log Rank — These results are using survival curve estimates to first positive urine toxicology for any opioid. The last observation carried forward (LOCF) was used to perform our survival event analyses; Cox Proportional Hazard = 2.4

ADVERSE EVENTS:
Time Frame: Adverse events were collected from week 1 to week 13.
Arm/Group | Memantine 30mg/Day + Buprenorphine | Memantine 15mg/Day + Buprenorphine | Memantine 0mg/Day + Buprenorphine
Serious Adverse Events (participants affected / at risk) | 0/27 | 0/24 | 0/29
Other Adverse Events (participants affected / at risk) | 18/27 | 15/24 | 23/29
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Memantine 30mg/Day + Buprenorphine (N=27) | Memantine 15mg/Day + Buprenorphine (N=24) | Memantine 0mg/Day + Buprenorphine (N=29)
Pain (Nervous system disorders) | 3 (5) | 3 (5) | 9 (15)
Upper Respiratory Intection (Respiratory, thoracic and mediastinal disorders) | 3 (5) | 1 (2) | 2 (4)
Nausea (Gastrointestinal disorders) | 2 (2) | 2 (2) | 4 (5)
Vivid Dreams (Psychiatric disorders) | 3 (3) | 2 (2) | 3 (3)
Constipation (Gastrointestinal disorders) | 4 (4) | 2 (2) | 1 (1)
Headache (Nervous system disorders) | 1 (1) | 3 (3) | 2 (2)
Drowsiness (Nervous system disorders) | 2 (2) | 2 (2) | 2 (2)

LIMITATIONS AND CAVEATS:
Rapid discontinuation of buprenorphine was associated with dropout that may have limited the statistical power to evaluate some variables. Memantine for 7 weeks may have been too short, and a longer exposure may have yielded better results.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No